CLINICAL TRIAL: NCT02969018
Title: A PHASE 2A, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE SAFETY AND EFFICACY OF PF-06700841 IN SUBJECTS WITH MODERATE TO SEVERE PLAQUE PSORIASIS
Brief Title: Study To Evaluate Safety And Efficacy Of PF-06700841 In Subjects With Moderate To Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7931004; 2016-004049-96 (EudraCT Number)
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Chronic Plaque Psoriasis
Keywords: plaque psoriasis
MeSH Terms: interventions — PF-06700841

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- PF-06700841 60 mg followed by 30 mg once daily (Experimental): 4 week induction with 60 mg PF-06700841 once daily, followed by 8 week chronic administration of 30 mg PF-06700841 once daily
  Interventions: Drug: PF-06700841
- PF-06700841 60 mg followed by 10 mg once daily (Experimental): 4 week induction with 60 mg PF-06700841 once daily, followed by 8 week chronic administration of 10 mg PF-06700841 once daily
  Interventions: Drug: PF-06700841
- PF-06700841 60mg once daily followed by 100mg once weekly (Experimental): 4 week induction with 60 mg PF-06700841 once daily, followed by 8 week chronic administration of 100 mg PF-06700841 once weekly
  Interventions: Drug: PF-06700841
- PF-06700841 60mg once daily followed by placebo once daily (Experimental): 4 week induction with 60 mg PF-06700841 once daily, followed by 8 week chronic administration of placebo once daily
  Interventions: Drug: PF-06700841
- PF-06700841 30mg once daily (Experimental): 4 week induction with 30 mg PF-06700841 once daily followed by 8 week chronic administration of 30 mg PF-06700841 once daily
  Interventions: Drug: PF-06700841
- PF-06700841 30mg once daily followed by 10mg once daily (Experimental): 4 week induction with 30 mg PF-06700841 once daily, followed by 8 week chronic administration of 10 mg PF-06700841 once daily
  Interventions: Drug: PF-06700841
- PF-06700841 30mg once daily followed by 100mg once weekly (Experimental): 4 week induction with 30 mg PF-06700841 once daily, followed by 8 week chronic administration of 100 mg PF-06700841 once weekly
  Interventions: Drug: PF-06700841
- Placebo (Placebo Comparator): 12 weeks once daily placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-06700841
  Arms: PF-06700841 30mg once daily; PF-06700841 30mg once daily followed by 100mg once weekly; PF-06700841 30mg once daily followed by 10mg once daily; PF-06700841 60 mg followed by 10 mg once daily; PF-06700841 60 mg followed by 30 mg once daily; PF-06700841 60mg once daily followed by 100mg once weekly; PF-06700841 60mg once daily followed by placebo once daily
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether PF-06700841 is safe and effective in the treatment of chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have had a diagnosis of plaque psoriasis (psoriasis vulgaris) for at least 6 months prior to Baseline/Day 1 (prior to first dose of study drug)
* Have a PASI score of 12 or greater AND a PGA score of 3 ("moderate") or 4 ("severe") at Baseline/Day 1 (prior to first dose of study drug)
* Have plaque-type psoriasis covering at least 10% of total body surface area (BSA) at Baseline/Day 1 (prior to first dose of study drug)
* Considered by dermatologist investigator to be a candidate for systemic therapy or phototherapy of psoriasis (either naïve or history of previous treatment)

Exclusion Criteria:

* Currently have non-plaque forms of psoriasis, eg, erythrodermic, guttate, or pustular psoriasis, with the exception of nail psoriasis which is allowed
* Have evidence of skin conditions (eg, eczema) at the time of screening or baseline visit that would interfere with the evaluation of psoriasis
* Cannot discontinue systemic therapies and/or topical therapies for the treatment of psoriasis and cannot discontinue phototherapy (UVB or PUVA)
* Have previously been treated with Secukinumab (Cosentyx), and Ixekizumab (Taltz).
* Have taken Apremilast (Otezla) within 3 months of first dose of study drug.
* Have undergone treatment with tofacitinib within 3 months of first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (30):
  - Northwest Arkansas Clinical Trials Center, PLLC/Hull Dermatology, PA, Rogers, Arkansas
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Emil A. Tanghetti, MD dba Center for Dermatology and Laser Surgery, Sacramento, California
  - Southern California Dermatology, Santa Ana, California
  - Tower Saint John's Imaging, Santa Monica, California
  - Clinical Science Institute, Santa Monica, California
  - Park Avenue Dermatology Administrative Annex, Orange Park, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Rose Radiology, Tampa, Florida
  - Forward Clinical Trials, Inc, Tampa, Florida
  - Dundee Dermatology, West Dundee, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dawes Fretzin Dermatology Group, LLC, Indianapolis, Indiana
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - The Rockefeller University, New York, New York
  - Skin Search of Rochester, Inc., Rochester, New York
  - Investigational Drug Services, UNC Hospitals, Chapel Hill, North Carolina
  - UNC Dermatology and Skin Cancer Center, Chapel Hill, North Carolina
  - UNC Clinical and Translation Research Center, Chapel Hill, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C, Tulsa, Oklahoma
  - Health Concepts, Rapid City, South Dakota
  - Center for Clinical Studies, Houston, Texas
  - Lee Medical Associates, PA, San Antonio, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Premier Clinical Research, Spokane, Washington
- Canada (8):
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Lynderm Research Inc, Markham, Ontario
  - Research by ICLS, Oakville, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - K.Papp Clinical Research Inc., Waterloo, Ontario
  - Centre de Recherche Dermatologique du Quebec metropolitain (CRDQ), Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Poland (6):
  - Centrum Medyczne Enel-Med Przychodnia Grunwaldzka, Gdansk
  - Centrum Badan Klinicznych PI-House Sp. z o.o., Gdansk
  - Dermoklinika Centrum Medyczne s.c. M.Kierstan, J. Narbutt, A. Lesiak, Lodz
  - NZOZ "Nasz Lekarz" - Praktyka Grupowa Lekarzy Rodzinnych z Przychodnia Specjalistyczna, Torun
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - WroMedica s.c., Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hughes JH, Qiu R, Banfield C, Dowty ME, Nicholas T. Population Pharmacokinetics of Oral Brepocitinib in Healthy Volunteers and Patients. Clin Pharmacol Drug Dev. 2022 Dec;11(12):1447-1456. doi: 10.1002/cpdd.1163. Epub 2022 Aug 31. PMID 36045513
- [Derived] Forman SB, Pariser DM, Poulin Y, Vincent MS, Gilbert SA, Kieras EM, Qiu R, Yu D, Papacharalambous J, Tehlirian C, Peeva E. TYK2/JAK1 Inhibitor PF-06700841 in Patients with Plaque Psoriasis: Phase IIa, Randomized, Double-Blind, Placebo-Controlled Trial. J Invest Dermatol. 2020 Dec;140(12):2359-2370.e5. doi: 10.1016/j.jid.2020.03.962. Epub 2020 Apr 18. PMID 32311398
- [Derived] Fensome A, Ambler CM, Arnold E, Banker ME, Brown MF, Chrencik J, Clark JD, Dowty ME, Efremov IV, Flick A, Gerstenberger BS, Gopalsamy A, Hayward MM, Hegen M, Hollingshead BD, Jussif J, Knafels JD, Limburg DC, Lin D, Lin TH, Pierce BS, Saiah E, Sharma R, Symanowicz PT, Telliez JB, Trujillo JI, Vajdos FF, Vincent F, Wan ZK, Xing L, Yang X, Yang X, Zhang L. Dual Inhibition of TYK2 and JAK1 for the Treatment of Autoimmune Diseases: Discovery of (( S)-2,2-Difluorocyclopropyl)((1 R,5 S)-3-(2-((1-methyl-1 H-pyrazol-4-yl)amino)pyrimidin-4-yl)-3,8-diazabicyclo[3.2.1]octan-8-yl)methanone (PF-06700841). J Med Chem. 2018 Oct 11;61(19):8597-8612. doi: 10.1021/acs.jmedchem.8b00917. Epub 2018 Aug 16. PMID 30113844
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7931004&StudyName=A+Phase+2a%2C+Randomized%2C+Double-blind%2C+Placebo-controlled+Study+To+Evaluate+Safety+And+Efficacy+Of+Pf-06700841+In+Subjects+With+Moderate+To+Severe+Plaque+Psoriasis

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD: Participants received 4-week induction of PF-06700841 60 mg QD (blinded tablets) followed by 8-week maintenance of PF-06700841 30 mg QD (blinded tablets).
- PF-06700841 60 mg QD Followed by 10 mg QD: Participants received 4-week induction of PF-06700841 60 mg QD (blinded tablets) followed by 8-week maintenance of PF-06700841 10 mg QD (blinded tablets).
- PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW): Participants received 4-week induction of PF-06700841 60 mg QD (blinded tablets) followed by 8-week maintenance of PF-06700841 100 mg QW (blinded tablets).
- PF-06700841 60 mg QD Followed by Placebo: Participants received 4-week induction of PF-06700841 60 mg QD (blinded tablets) followed by 8-week maintenance of matching placebo QD (blinded tablets).
- PF-06700841 30 mg QD: Participants received 12 weeks of blinded PF-06700841 30 mg QD tablets.
- PF-06700841 30 mg QD Followed by 10 mg QD: Participants received 4-week induction of PF-06700841 30 mg QD (blinded tablets) followed by 8-week maintenance of PF-06700841 10 mg QD (blinded tablets).
- PF-06700841 30 mg QD Followed by 100 mg QW: Participants received 4-week induction of PF-06700841 30 mg QD (blinded tablets) followed by 8-week maintenance of PF-06700841 100 mg QW (blinded tablets).
- Placebo: Participants received 12 weeks of blinded matching placebo QD tablets.
Period: Overall Study
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Started | 25 | 29 | 26 | 25 | 29 | 25 | 30 | 23
Completed | 21 | 21 | 20 | 20 | 27 | 17 | 22 | 16
Not Completed | 4 | 8 | 6 | 5 | 2 | 8 | 8 | 7
Not completed — Adverse Event | 2 | 4 | 1 | 2 | 0 | 1 | 2 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 2 | 0 | 1 | 1 | 0 | 1
Not completed — No Longer Meets Eligibility Criteria | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Non-Compliance With Study Drug | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 1 | 0 | 4 | 4 | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of PF-06700841 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo | Total
Number analyzed (Participants) | 25 | 29 | 26 | 25 | 29 | 25 | 30 | 23 | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (14.69) | 44.6 (13.71) | 45.5 (12.93) | 48.4 (15.47) | 44.2 (10.92) | 44.0 (11.56) | 43.2 (12.28) | 50.3 (12.23) | 46.0 (13.04)
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 8 | 14 | 10 | 8 | 14 | 12 | 14 | 8 | 88
  45-64 Years | 14 | 13 | 14 | 13 | 14 | 13 | 16 | 12 | 109
  >=65 Years | 3 | 2 | 2 | 4 | 1 | 0 | 0 | 3 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 14 | 4 | 10 | 8 | 7 | 4 | 64
  Male | 16 | 21 | 12 | 21 | 19 | 17 | 23 | 19 | 148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 4 | 2 | 6 | 5 | 4 | 4 | 33
  Not Hispanic or Latino | 21 | 25 | 22 | 23 | 23 | 20 | 26 | 19 | 179
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 27 | 23 | 24 | 27 | 22 | 25 | 19 | 189
  Black or African American | 3 | 0 | 3 | 0 | 1 | 1 | 1 | 2 | 11
  Asian | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 4
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Other | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 12
Description: The PASI quantifies the severity of a participant's psoriasis based on both lesion severity and the percentage of body surface area (BSA) affected. In each area, the sum of the severity rating scores for erythema, induration and scaling is multiplied by the score representing the percentage of this area involved by psoriasis, multiplied by a weighting factor (head 0.1; upper limbs 0.2; trunk 0.3; lower limbs 0.4). The sum of the numbers obtained for each of the four body areas is the PASI. The PASI score can vary in increments of 0.1 units from 0.0 to 72.0, with higher scores representing increasing severity of psoriasis.
Time Frame: Baseline (Day 1 pre-dose), Week 12
Population: All randomized participants who received at least 1 dose of investigational product (PF-06700841 or placebo) and had observed PASI data for Week 12.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Number analyzed (Participants) | 22 | 21 | 21 | 21 | 27 | 19 | 25 | 17
units on a scale | -15.85 [-18.31 to -13.39] | -10.56 [-12.96 to -8.16] | -14.28 [-16.75 to -11.81] | -10.14 [-12.62 to -7.66] | -17.28 [-19.55 to -15.02] | -13.27 [-15.78 to -10.76] | -11.88 [-14.16 to -9.59] | -7.21 [-9.96 to -4.46]
Statistical Analysis 1: Comparison: PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD vs Placebo; Test type: Other; p = 0.0005, Mixed Models Analysis — Hochberg adjusted p-value; Least Squares Mean Difference = -8.64, 90% CI 2-sided [-12.33 to -4.95], Standard Error of Mean 2.232
Statistical Analysis 2: Comparison: PF-06700841 60 mg QD Followed by 10 mg QD vs Placebo; Test type: Other; p = 0.0963, Mixed Models Analysis — Hochberg adjusted p-value; Least Squares Mean Difference = -3.34, 90% CI 2-sided [-6.99 to 0.30], Standard Error of Mean 2.206
Statistical Analysis 3: Comparison: PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) vs Placebo; Test type: Other; p = 0.0046, Mixed Models Analysis — Hochberg adjusted p-value; Least Squares Mean Difference = -7.07, 90% CI 2-sided [-10.76 to -3.37], Standard Error of Mean 2.233
Statistical Analysis 4: Comparison: PF-06700841 60 mg QD Followed by Placebo vs Placebo; Test type: Other; p = 0.0963, Mixed Models Analysis — Hochberg adjusted p-value; Least Squares Mean Difference = -2.93, 90% CI 2-sided [-6.63 to 0.77], Standard Error of Mean 2.238
Statistical Analysis 5: Comparison: PF-06700841 30 mg QD vs Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis — Hochberg adjusted p-value; Least Squares Mean Difference = -10.07, 90% CI 2-sided [-13.63 to -6.51], Standard Error of Mean 2.152
Statistical Analysis 6: Comparison: PF-06700841 30 mg QD Followed by 10 mg QD vs Placebo; Test type: Other; p = 0.0158, Mixed Models Analysis — Hochberg adjusted p-value; Least Squares Mean Difference = -6.06, 90% CI 2-sided [-9.79 to -2.33], Standard Error of Mean 2.255
Statistical Analysis 7: Comparison: PF-06700841 30 mg QD Followed by 100 mg QW vs Placebo; Test type: Other; p = 0.0488, Mixed Models Analysis — Hochberg adjusted p-value; Least Squares Mean Difference = -4.66, 90% CI 2-sided [-8.24 to -1.09], Standard Error of Mean 2.163

2. Secondary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index 75 (PASI75) Response at Week 12
Description: A PASI75 response is a 75% or greater reduction from baseline in PASI score. The PASI score can vary in increments of 0.1 units from 0.0 to 72.0, with higher scores representing increasing severity of psoriasis.
Time Frame: Week 12
Population: All participants who received at least 1 dose of investigational product (PF-06700841 or placebo) with PASI data at Week 12 after non-responder imputation applied.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Number analyzed (Participants) | 25 | 29 | 26 | 25 | 29 | 25 | 30 | 23
percentage of participants | 60.0 [41.68 to 76.44] | 24.1 [11.92 to 40.60] | 57.7 [39.84 to 74.16] | 24.0 [11.01 to 41.95] | 86.2 [71.16 to 95.15] | 24.0 [11.01 to 41.95] | 36.7 [22.11 to 53.31] | 13.0 [3.65 to 30.36]
Statistical Analysis 1: Comparison: PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD vs Placebo; Test type: Other; Odds Ratio (OR) = 10.00, 90% CI 2-sided [2.95 to 33.87]; Logistic regression
Statistical Analysis 2: Comparison: PF-06700841 60 mg QD Followed by 10 mg QD vs Placebo; Test type: Other; Odds Ratio (OR) = 2.12, 90% CI 2-sided [0.61 to 7.36]; Logistic regression
Statistical Analysis 3: Comparison: PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) vs Placebo; Test type: Other; Odds Ratio (OR) = 9.09, 90% CI 2-sided [2.71 to 30.48]; Logistic regression
Statistical Analysis 4: Comparison: PF-06700841 60 mg QD Followed by Placebo vs Placebo; Test type: Other; Odds Ratio (OR) = 2.11, 90% CI 2-sided [0.59 to 7.55]; Logistic regression
Statistical Analysis 5: Comparison: PF-06700841 30 mg QD vs Placebo; Test type: Other; Odds Ratio (OR) = 41.67, 90% CI 2-sided [10.80 to 160.68]; Logistic regression
Statistical Analysis 6: Comparison: PF-06700841 30 mg QD Followed by 10 mg QD vs Placebo; Test type: Other; Odds Ratio (OR) = 2.11, 90% CI 2-sided [0.59 to 7.55]; Logistic regression
Statistical Analysis 7: Comparison: PF-06700841 30 mg QD Followed by 100 mg QW vs Placebo; Test type: Other; Odds Ratio (OR) = 3.86, 90% CI 2-sided [1.17 to 12.74]; Logistic regression

3. Secondary Outcome: Change From Baseline in PASI Scores at Week 4 by Induction Dose
Description: Change from baseline in PASI scores at Week 4 was presented by induction dose (ie, PF-06700841 60 mg QD, 30 mg QD, and placebo). The PASI score can vary in increments of 0.1 units from 0.0 to 72.0, with higher scores representing increasing severity of psoriasis.
Time Frame: Baseline (Day 1 pre-dose), Week 4
Population: All participants who received at least 1 dose of investigational product (PF-06700841 or placebo) and had observed PASI data at Week 4.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Groups:
- PF-06700841 60 mg QD as the Induction Dose: Participants received PF-06700841 60 mg QD as the induction dose.
- PF-06700841 30 mg QD as the Induction Dose: Participants received PF-06700841 30 mg QD as the induction dose.
- Placebo as the Induction Dose: Participants received matching placebo QD as the induction dose.
Arm/Group | PF-06700841 60 mg QD as the Induction Dose | PF-06700841 30 mg QD as the Induction Dose | Placebo as the Induction Dose
Number analyzed (Participants) | 100 | 81 | 21
units on a scale | -13.17 [-14.20 to -12.15] | -12.16 [-13.31 to -11.02] | -4.17 [-6.38 to -1.97]
Statistical Analysis 1: Comparison: PF-06700841 60 mg QD as the Induction Dose vs Placebo as the Induction Dose; Test type: Other; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -9.00, 90% CI 2-sided [-11.43 to -6.57], Standard Error of Mean 1.470
Statistical Analysis 2: Comparison: PF-06700841 30 mg QD as the Induction Dose vs Placebo as the Induction Dose; Test type: Other; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -7.99, 90% CI 2-sided [-10.48 to -5.51], Standard Error of Mean 1.502

4. Secondary Outcome: Percentage of Participants Achieving PASI75 Responses at Weeks 1, 2, 4, 6, 8, 10, 14, 16
Description: as for outcome 2
Time Frame: Weeks 1, 2, 4, 6, 8, 10, 14, 16
Population: All participants who received at least 1 dose of investigational product (PF-06700841 or placebo) with PASI data for each specified time point after non-responder imputation applied.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Number analyzed (Participants) | 25 | 29 | 26 | 25 | 29 | 25 | 30 | 23
percentage of participants
  Week 1 | 0 [0.00 to 11.29] | 6.9 [1.24 to 20.16] | 7.7 [1.38 to 22.29] | 4.0 [0.20 to 17.61] | 0 [0.00 to 9.81] | 4.0 [0.20 to 17.61] | 0 [0.00 to 9.50] | 0 [0.00 to 12.21]
  Week 2 | 8.0 [1.44 to 23.10] | 13.8 [4.85 to 28.84] | 26.9 [13.38 to 44.68] | 12.0 [3.35 to 28.17] | 3.4 [0.18 to 15.34] | 8.0 [1.44 to 23.10] | 0 [0.00 to 9.50] | 0 [0.00 to 12.21]
  Week 4 | 24.0 [11.01 to 41.95] | 41.4 [25.89 to 58.25] | 61.5 [43.57 to 77.43] | 36.0 [20.24 to 54.39] | 27.6 [14.53 to 44.29] | 24.0 [11.01 to 41.95] | 36.7 [22.11 to 53.31] | 0 [0.00 to 12.21]
  Week 6 | 44.0 [26.99 to 62.14] | 41.4 [25.89 to 58.25] | 65.4 [47.38 to 80.60] | 36.0 [20.24 to 54.39] | 51.7 [35.20 to 67.97] | 28.0 [13.95 to 46.22] | 26.7 [14.02 to 42.99] | 8.7 [1.57 to 24.92]
  Week 8 | 60.0 [41.68 to 76.44] | 37.9 [22.93 to 54.88] | 65.4 [47.38 to 80.60] | 32.0 [17.03 to 50.36] | 65.5 [48.57 to 79.95] | 20.0 [8.23 to 37.54] | 40.0 [24.95 to 56.61] | 8.7 [1.57 to 24.92]
  Week 10 | 48.0 [30.51 to 65.86] | 24.1 [11.92 to 40.60] | 61.5 [43.57 to 77.43] | 32.0 [17.03 to 50.36] | 72.4 [55.71 to 85.47] | 28.0 [13.95 to 46.22] | 46.7 [30.85 to 63.01] | 13.0 [3.65 to 30.36]
  Week 14 | 48.0 [30.51 to 65.86] | 17.2 [7.05 to 32.89] | 34.6 [19.40 to 52.62] | 16.0 [5.66 to 32.96] | 75.9 [59.40 to 88.08] | 16.0 [5.66 to 32.96] | 16.7 [6.81 to 31.90] | 8.7 [1.57 to 24.92]
  Week 16 | 36.0 [20.24 to 54.39] | 10.3 [2.88 to 24.61] | 30.8 [16.33 to 48.70] | 20.0 [8.23 to 37.54] | 58.6 [41.75 to 74.11] | 12.0 [3.35 to 28.17] | 16.7 [6.81 to 31.90] | 8.7 [1.57 to 24.92]

5. Secondary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index 50 (PASI50) Response at Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16
Description: A PASI50 response is a 50% or greater reduction from baseline in PASI score. The PASI score can vary in increments of 0.1 units from 0.0 to 72.0, with higher scores representing increasing severity of psoriasis.
Time Frame: Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Number analyzed (Participants) | 25 | 29 | 26 | 25 | 29 | 25 | 30 | 23
percentage of participants
  Week 1 | 12.0 [3.35 to 28.17] | 13.8 [4.85 to 28.84] | 19.2 [7.90 to 36.26] | 20.0 [8.23 to 37.54] | 10.3 [2.88 to 24.61] | 8.0 [1.44 to 23.10] | 3.3 [0.17 to 14.86] | 0 [0.00 to 12.21]
  Week 2 | 44.0 [26.99 to 62.14] | 37.9 [22.93 to 54.88] | 46.2 [29.21 to 63.79] | 32.0 [17.03 to 50.36] | 41.4 [25.89 to 58.25] | 20.0 [8.23 to 37.54] | 33.3 [19.33 to 49.94] | 0 [0.00 to 12.21]
  Week 4 | 60.0 [41.68 to 76.44] | 69.0 [52.10 to 82.75] | 69.2 [51.30 to 83.67] | 68.0 [49.64 to 82.97] | 69.0 [52.10 to 82.75] | 60.0 [41.68 to 76.44] | 66.7 [50.06 to 80.67] | 13.0 [3.65 to 30.36]
  Week 6 | 72.0 [53.78 to 86.05] | 62.1 [45.12 to 77.07] | 73.1 [55.32 to 86.62] | 68.0 [49.64 to 82.97] | 82.8 [67.11 to 92.95] | 60.0 [41.68 to 76.44] | 63.3 [46.69 to 77.89] | 26.1 [12.02 to 45.10]
  Week 8 | 72.0 [53.78 to 86.05] | 55.2 [38.44 to 71.07] | 73.1 [55.32 to 86.62] | 52.0 [34.14 to 69.49] | 86.2 [71.16 to 95.15] | 56.0 [37.86 to 73.01] | 63.3 [46.69 to 77.89] | 17.4 [6.17 to 35.49]
  Week 10 | 68.0 [49.64 to 82.97] | 44.8 [28.93 to 61.56] | 73.1 [55.32 to 86.62] | 48.0 [30.51 to 65.86] | 86.2 [71.16 to 95.15] | 48.0 [30.51 to 65.86] | 56.7 [40.16 to 72.13] | 17.4 [6.17 to 35.49]
  Week 12 | 68.0 [49.64 to 82.97] | 44.8 [28.93 to 61.56] | 69.2 [51.30 to 83.67] | 52.0 [34.14 to 69.49] | 89.7 [75.39 to 97.12] | 48.0 [30.51 to 65.86] | 53.3 [36.99 to 69.15] | 21.7 [8.98 to 40.39]
  Week 14 | 64.0 [45.61 to 79.76] | 44.8 [28.93 to 61.56] | 61.5 [43.57 to 77.43] | 48.0 [30.51 to 65.86] | 89.7 [75.39 to 97.12] | 36.0 [20.24 to 54.39] | 36.7 [22.11 to 53.31] | 26.1 [12.02 to 45.10]
  Week 16 | 60.0 [41.68 to 76.44] | 34.5 [20.05 to 51.43] | 53.8 [36.21 to 70.79] | 40.0 [23.56 to 58.32] | 79.3 [63.20 to 90.58] | 40.0 [23.56 to 58.32] | 36.7 [22.11 to 53.31] | 21.7 [8.98 to 40.39]

6. Secondary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index 90 (PASI90) Response at Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16
Description: A PASI90 response is a 90% or greater reduction from baseline in PASI score. The PASI score can vary in increments of 0.1 units from 0.0 to 72.0, with higher scores representing increasing severity of psoriasis.
Time Frame: Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Number analyzed (Participants) | 25 | 29 | 26 | 25 | 29 | 25 | 30 | 23
percentage of participants
  Week 1 | 0 [0.00 to 11.29] | 3.4 [0.18 to 15.34] | 0 [0.00 to 10.88] | 0 [0.00 to 11.29] | 0 [0.00 to 9.81] | 0 [0.00 to 11.29] | 0 [0.00 to 9.50] | 0 [0.00 to 12.21]
  Week 2 | 0 [0.00 to 11.29] | 3.4 [0.18 to 15.34] | 7.7 [1.38 to 22.29] | 0 [0.00 to 11.29] | 0 [0.00 to 9.81] | 0 [0.00 to 11.29] | 0 [0.00 to 9.50] | 0 [0.00 to 12.21]
  Week 4 | 12.0 [3.35 to 28.17] | 20.7 [9.42 to 36.80] | 42.3 [25.84 to 60.16] | 16.0 [5.66 to 32.96] | 6.9 [1.24 to 20.16] | 8.0 [1.44 to 23.10] | 3.3 [0.17 to 14.86] | 0 [0.00 to 12.21]
  Week 6 | 16.0 [5.66 to 32.96] | 20.7 [9.42 to 36.80] | 26.9 [13.38 to 44.68] | 12.0 [3.35 to 28.17] | 24.1 [11.92 to 40.60] | 8.0 [1.44 to 23.10] | 20.0 [9.09 to 35.70] | 0 [0.00 to 12.21]
  Week 8 | 24.0 [11.01 to 41.95] | 17.2 [7.05 to 32.89] | 30.8 [16.33 to 48.70] | 8.0 [1.44 to 23.10] | 34.5 [20.05 to 51.43] | 4.0 [0.20 to 17.61] | 16.7 [6.81 to 31.90] | 0 [0.00 to 12.21]
  Week 10 | 28.0 [13.95 to 46.22] | 17.2 [7.05 to 32.89] | 26.9 [13.38 to 44.68] | 8.0 [1.44 to 23.10] | 34.5 [20.05 to 51.43] | 8.0 [1.44 to 23.10] | 13.3 [4.69 to 27.96] | 4.3 [0.22 to 19.02]
  Week 12 | 36.0 [20.24 to 54.39] | 13.8 [4.85 to 28.84] | 26.9 [13.38 to 44.68] | 8.0 [1.44 to 23.10] | 51.7 [35.20 to 67.97] | 8.0 [1.44 to 23.10] | 10.0 [2.78 to 23.86] | 4.3 [0.22 to 19.02]
  Week 14 | 28.0 [13.95 to 46.22] | 13.8 [4.85 to 28.84] | 11.5 [3.22 to 27.19] | 8.0 [1.44 to 23.10] | 37.9 [22.93 to 54.88] | 4.0 [0.20 to 17.61] | 13.3 [4.69 to 27.96] | 4.3 [0.22 to 19.02]
  Week 16 | 20.0 [8.23 to 37.54] | 3.4 [0.18 to 15.34] | 15.4 [5.43 to 31.82] | 4.0 [0.20 to 17.61] | 27.6 [14.53 to 44.29] | 8.0 [1.44 to 23.10] | 10.0 [2.78 to 23.86] | 4.3 [0.22 to 19.02]

7. Secondary Outcome: Change From Baseline in PASI Scores at Weeks 1, 2, 4, 6, 8, 10, 14, 16
Description: The PASI score can vary in increments of 0.1 units from 0.0 to 72.0, with higher scores representing increasing severity of psoriasis.
Time Frame: Baseline (Day 1 pre-dose), Weeks 1, 2, 4, 6, 8, 10, 14, 16
Population: "Number of participants analyzed" represents all participants who received at least 1 dose of investigational product (PF-06700841 or placebo). "Number analyzed" represents all participants who received at least 1 dose of investigational product (PF-06700841 or placebo) and had observed PASI data for each specified time point.
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Number analyzed (Participants) | 25 | 29 | 26 | 25 | 29 | 25 | 30 | 23
units on a scale
  Week 1: number analyzed (Participants) | 25 | 29 | 24 | 25 | 28 | 25 | 30 | 23
  Week 1 | -5.74 [-7.61 to -3.86] | -4.60 [-6.06 to -3.14] | -5.85 [-7.62 to -4.08] | -5.37 [-7.59 to -3.15] | -3.97 [-5.00 to -2.95] | -4.41 [-6.18 to -2.64] | -3.46 [-4.64 to -2.28] | -1.35 [-2.03 to -0.66]
  Week 2: number analyzed (Participants) | 24 | 28 | 24 | 24 | 28 | 25 | 30 | 21
  Week 2 | -9.44 [-11.74 to -7.15] | -8.35 [-10.07 to -6.63] | -10.79 [-13.05 to -8.52] | -9.49 [-12.40 to -6.58] | -7.86 [-9.38 to -6.35] | -7.79 [-9.79 to -5.79] | -7.93 [-9.64 to -6.22] | -2.28 [-3.21 to -1.36]
  Week 4: number analyzed (Participants) | 23 | 28 | 25 | 24 | 28 | 25 | 28 | 21
  Week 4 | -12.85 [-15.76 to -9.94] | -12.19 [-14.57 to -9.81] | -14.11 [-16.37 to -11.86] | -13.91 [-16.98 to -10.85] | -11.72 [-13.61 to -9.83] | -12.88 [-15.49 to -10.27] | -13.06 [-15.58 to -10.53] | -4.02 [-6.04 to -2.00]
  Week 6: number analyzed (Participants) | 23 | 25 | 24 | 23 | 28 | 24 | 27 | 19
  Week 6 | -15.00 [-18.30 to -11.71] | -12.12 [-14.53 to -9.71] | -15.00 [-17.35 to -12.66] | -13.85 [-16.62 to -11.08] | -14.30 [-16.24 to -12.36] | -14.33 [-17.47 to -11.19] | -14.17 [-16.92 to -11.41] | -5.52 [-7.58 to -3.45]
  Week 8: number analyzed (Participants) | 23 | 24 | 22 | 22 | 27 | 21 | 27 | 17
  Week 8 | -15.94 [-19.40 to -12.49] | -11.09 [-12.90 to -9.27] | -14.97 [-17.66 to -12.27] | -12.87 [-15.69 to -10.04] | -15.82 [-17.81 to -13.84] | -14.27 [-17.51 to -11.03] | -13.83 [-16.79 to -10.87] | -6.56 [-8.61 to -4.51]
  Week 10: number analyzed (Participants) | 21 | 22 | 22 | 23 | 26 | 21 | 27 | 17
  Week 10 | -16.54 [-20.54 to -12.54] | -9.89 [-12.16 to -7.61] | -15.52 [-18.09 to -12.96] | -11.64 [-14.92 to -8.37] | -16.65 [-18.64 to -14.66] | -14.98 [-18.43 to -11.53] | -12.97 [-16.19 to -9.74] | -6.78 [-9.20 to -4.37]
  Week 14: number analyzed (Participants) | 21 | 21 | 21 | 22 | 27 | 19 | 24 | 16
  Week 14 | -15.47 [-19.88 to -11.06] | -8.11 [-10.69 to -5.53] | -13.31 [-16.73 to -9.89] | -9.45 [-12.96 to -5.94] | -16.14 [-18.16 to -14.12] | -10.44 [-13.33 to -7.55] | -11.03 [-14.61 to -7.44] | -6.98 [-9.81 to -4.14]
  Week 16: number analyzed (Participants) | 21 | 21 | 20 | 21 | 26 | 18 | 23 | 16
  Week 16 | -14.16 [-18.68 to -9.64] | -6.59 [-9.09 to -4.09] | -13.00 [-16.60 to -9.40] | -7.83 [-11.56 to -4.11] | -14.38 [-16.74 to -12.01] | -9.62 [-13.08 to -6.16] | -9.13 [-13.94 to -4.33] | -6.76 [-9.80 to -3.72]

8. Secondary Outcome: Percent Change From Baseline in PASI Scores at Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16
Description: as for outcome 7
Time Frame: Baseline (Day 1 pre-dose), Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16
Population: as for outcome 7
Measure: Mean (90% Confidence Interval); unit: percent change
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Number analyzed (Participants) | 25 | 29 | 26 | 25 | 29 | 25 | 30 | 23
percent change
  Week 1: number analyzed (Participants) | 25 | 29 | 24 | 25 | 28 | 25 | 30 | 23
  Week 1 | -26.70 [-33.80 to -19.60] | -24.66 [-33.24 to -16.08] | -30.25 [-39.07 to -21.44] | -23.33 [-30.84 to -15.82] | -20.92 [-26.82 to -15.01] | -17.50 [-23.91 to -11.10] | -15.42 [-20.68 to -10.16] | -6.90 [-10.50 to -3.30]
  Week 2: number analyzed (Participants) | 24 | 28 | 24 | 24 | 28 | 25 | 30 | 21
  Week 2 | -43.66 [-52.81 to -34.52] | -44.17 [-52.75 to -35.59] | -54.27 [-64.17 to -44.36] | -42.58 [-51.17 to -33.98] | -40.89 [-47.94 to -33.83] | -32.46 [-39.75 to -25.16] | -35.89 [-42.69 to -29.09] | -12.81 [-18.29 to -7.33]
  Week 4: number analyzed (Participants) | 23 | 28 | 25 | 24 | 28 | 25 | 28 | 21
  Week 4 | -57.16 [-67.35 to -46.97] | -63.02 [-72.12 to -53.91] | -72.41 [-82.31 to -62.51] | -64.71 [-72.81 to -56.61] | -60.76 [-68.38 to -53.14] | -53.93 [-62.59 to -45.28] | -58.99 [-67.94 to -50.03] | -25.17 [-34.24 to -16.09]
  Week 6: number analyzed (Participants) | 23 | 25 | 24 | 23 | 28 | 24 | 27 | 19
  Week 6 | -66.07 [-76.06 to -56.08] | -63.31 [-73.99 to -52.62] | -75.96 [-84.68 to -67.25] | -65.06 [-74.15 to -55.97] | -73.91 [-80.62 to -67.19] | -58.57 [-66.76 to -50.37] | -63.17 [-72.37 to -53.96] | -33.49 [-44.16 to -22.83]
  Week 8: number analyzed (Participants) | 23 | 24 | 22 | 22 | 27 | 21 | 27 | 17
  Week 8 | -70.11 [-80.95 to -59.27] | -62.25 [-72.42 to -52.07] | -77.05 [-86.69 to -67.41] | -59.88 [-69.78 to -49.97] | -81.04 [-86.69 to -75.40] | -58.32 [-66.39 to -50.25] | -61.38 [-71.80 to -50.96] | -37.76 [-47.73 to -27.80]
  Week 10: number analyzed (Participants) | 21 | 22 | 22 | 23 | 26 | 21 | 27 | 17
  Week 10 | -70.72 [-83.32 to -58.12] | -57.55 [-69.11 to -46.00] | -78.46 [-85.82 to -71.09] | -53.81 [-64.41 to -43.22] | -84.82 [-89.50 to -80.15] | -61.23 [-69.29 to -53.17] | -57.24 [-68.80 to -45.69] | -39.68 [-50.92 to -28.44]
  Week 12: number analyzed (Participants) | 22 | 21 | 21 | 21 | 27 | 19 | 25 | 17
  Week 12 | -71.94 [-84.67 to -59.21] | -58.52 [-69.38 to -47.67] | -74.42 [-84.98 to -63.87] | -51.49 [-63.21 to -39.78] | -88.68 [-93.13 to -84.22] | -57.81 [-68.52 to -47.10] | -58.57 [-70.05 to -47.09] | -40.27 [-52.68 to -27.86]
  Week 14: number analyzed (Participants) | 21 | 21 | 21 | 22 | 27 | 19 | 24 | 16
  Week 14 | -64.15 [-78.24 to -50.05] | -47.87 [-62.17 to -33.56] | -63.20 [-74.36 to -52.05] | -44.30 [-57.51 to -31.09] | -83.39 [-89.74 to -77.04] | -47.84 [-60.18 to -35.49] | -47.52 [-59.86 to -35.18] | -39.48 [-52.09 to -26.88]
  Week 16: number analyzed (Participants) | 21 | 21 | 20 | 21 | 26 | 18 | 23 | 16
  Week 16 | -57.28 [-72.02 to -42.54] | -38.48 [-51.85 to -25.10] | -60.56 [-72.71 to -48.42] | -36.63 [-51.43 to -21.83] | -74.18 [-83.22 to -65.15] | -44.58 [-58.96 to -30.19] | -42.29 [-59.96 to -24.63] | -38.79 [-51.92 to -25.66]

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE (non-serious and serious) was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening (immediate risk of death); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; or an important medical event. Any such events with initial onset or increasing in severity after the first dose of study treatment were counted as treatment-emergent.
Time Frame: From first dose of study treatment (Day 1) up to Week 20
Population: All participants who received at least 1 dose of investigational product (PF-06700841 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Number analyzed (Participants) | 25 | 29 | 26 | 25 | 29 | 25 | 30 | 23
Participants
  Treatment-emergent AEs | 19 | 21 | 18 | 18 | 21 | 16 | 23 | 13
  Treatment-emergent SAEs | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Who Discontinued From the Study Due to Treatment-Emergent AEs
Description: The number of participants who discontinued from the study due to treatment-emergent AEs is presented. Note for data reported under this Outcome Measure: Per sponsor reporting standard, pregnancy was counted as AE for AE data tables while it was counted separately in the disposition data table (Participant Flow Module).
Time Frame: From first dose of study treatment (Day 1) up to Week 20
Population: All participants who received at least 1 dose of investigational product (PF-06700841 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Number analyzed (Participants) | 25 | 29 | 26 | 25 | 29 | 25 | 30 | 23
Participants | 2 | 4 | 1 | 2 | 0 | 2 | 2 | 0

11. Secondary Outcome: Change From Baseline in Blood Lipid Level at Weeks 4 and 12
Description: Lipid panel included low density lipoprotein (LDL) cholesterol, high density lipoprotein (HDL) cholesterol, total cholesterol, and triglycerides.
Time Frame: Baseline (Day 1 pre-dose), Weeks 4 and 12
Population: "Number of participants analyzed" represents all participants who received at least 1 dose of investigational product (PF-06700841 or placebo). "Number analyzed" represents all participants who received at least 1 dose of investigational product (PF-06700841 or placebo) and had data for each specified category.
Measure: Mean (90% Confidence Interval); unit: milligram per deciliter (mg/dL)
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Number analyzed (Participants) | 25 | 29 | 26 | 25 | 29 | 25 | 30 | 23
milligram per deciliter (mg/dL)
  LDL Cholesterol, Week 4: number analyzed (Participants) | 22 | 26 | 21 | 24 | 23 | 24 | 25 | 18
  LDL Cholesterol, Week 4 | 15.91 [7.95 to 23.86] | 11.27 [4.31 to 18.23] | 15.00 [-0.63 to 30.63] | 15.88 [6.63 to 25.12] | 8.96 [0.99 to 16.92] | -2.21 [-11.04 to 6.63] | 7.60 [-4.39 to 19.59] | -6.28 [-10.56 to -2.00]
  LDL Cholesterol, Week 12: number analyzed (Participants) | 21 | 20 | 19 | 20 | 20 | 18 | 22 | 15
  LDL Cholesterol, Week 12 | 8.71 [1.04 to 16.39] | 6.00 [-4.73 to 16.73] | -0.74 [-11.67 to 10.20] | 6.85 [-2.06 to 15.76] | 14.10 [6.63 to 21.57] | -5.33 [-18.24 to 7.57] | 3.95 [-7.79 to 15.70] | -4.00 [-9.71 to 1.71]
  HDL Cholesterol, Week 4: number analyzed (Participants) | 23 | 28 | 25 | 24 | 28 | 25 | 28 | 19
  HDL Cholesterol, Week 4 | 12.09 [8.07 to 16.11] | 9.14 [5.84 to 12.45] | 10.92 [7.38 to 14.46] | 8.58 [5.84 to 11.33] | 6.36 [3.91 to 8.80] | 6.76 [2.93 to 10.59] | 9.39 [7.03 to 11.75] | 0.00 [-5.14 to 5.14]
  HDL Cholesterol, Week 12: number analyzed (Participants) | 22 | 21 | 21 | 21 | 27 | 19 | 24 | 15
  HDL Cholesterol, Week 12 | 5.00 [1.29 to 8.71] | 5.48 [1.66 to 9.29] | 2.48 [-0.31 to 5.26] | -0.24 [-2.55 to 2.08] | 4.74 [1.30 to 8.18] | 4.37 [1.04 to 7.70] | 2.88 [-0.24 to 5.99] | -2.73 [-6.32 to 0.85]
  Total Cholesterol, Week 4: number analyzed (Participants) | 23 | 28 | 25 | 24 | 28 | 25 | 28 | 19
  Total Cholesterol, Week 4 | 34.39 [24.01 to 44.77] | 29.46 [18.68 to 40.25] | 31.32 [15.20 to 47.44] | 26.33 [15.85 to 36.82] | 15.14 [-0.16 to 30.45] | 10.36 [-1.70 to 22.42] | 14.00 [0.14 to 27.86] | -4.42 [-10.90 to 2.06]
  Total Cholesterol, Week 12: number analyzed (Participants) | 22 | 21 | 21 | 21 | 27 | 19 | 24 | 15
  Total Cholesterol, Week 12 | 19.50 [9.95 to 29.05] | 15.67 [2.74 to 28.59] | -1.86 [-13.78 to 10.07] | 7.05 [-3.25 to 17.35] | 20.37 [3.06 to 37.68] | 0.68 [-14.51 to 15.87] | 4.33 [-8.86 to 17.53] | -6.40 [-13.68 to 0.88]
  Triglycerides, Week 4: number analyzed (Participants) | 23 | 28 | 25 | 24 | 28 | 25 | 28 | 19
  Triglycerides, Week 4 | 34.74 [-8.43 to 77.91] | 29.68 [10.42 to 48.94] | 8.04 [-20.07 to 36.15] | 8.92 [-21.83 to 39.66] | -65.11 [-204.94 to 74.72] | 19.60 [-3.04 to 42.24] | -59.75 [-157.79 to 38.29] | 15.26 [-11.07 to 41.60]
  Triglycerides, Week 12: number analyzed (Participants) | 22 | 21 | 21 | 21 | 27 | 19 | 24 | 15
  Triglycerides, Week 12 | 27.86 [-4.68 to 60.41] | 48.33 [-32.67 to 129.34] | -85.00 [-213.81 to 43.81] | 2.67 [-27.36 to 32.70] | -18.96 [-198.51 to 160.59] | 6.32 [-19.21 to 31.84] | -67.79 [-185.53 to 49.95] | 1.87 [-24.28 to 28.01]

12. Secondary Outcome: Number of Participants With Any Post-Baseline Laboratory Test Abnormalities
Description: Following laboratory parameters were assessed against pre-defined abnormality criteria: hematology (hemoglobin, hematocrit, erythrocytes, reticulocytes, platelets, leukocytes, lymphocytes, neutrophils, basophils, eosinophils, monocytes, activated partial thromboplastin time, prothrombin time [PT], PT/international normalized ratio; chemistry (total bilirubin, direct bilirubin, aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase, alkaline phosphatase, protein, albumin, urea nitrogen, creatinine, urate, total cholesterol, LDL and HDL cholesterol, triglycerides, calcium, sodium, potassium, chloride, bicarbonate, glucose, creatine kinase, Cystatin C, glomerular filtration rate; urinalysis (pH, urine glucose, ketones, urine protein, urine hemoglobin, nitrites, leukocyte esterase, urine erythrocytes, urine leukocytes, hyaline casts, bacteria, choriogonadotropin beta).
Time Frame: From first dose of study treatment (Day 1) up to Week 16
Population: All participants who received at least 1 dose of investigational product (PF-06700841 or placebo) and had post-baseline laboratory data.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Number analyzed (Participants) | 25 | 29 | 25 | 25 | 28 | 25 | 30 | 23
Participants | 17 | 20 | 20 | 16 | 21 | 20 | 18 | 11

13. Secondary Outcome: Number of Participants With Post-Baseline Vital Sign Abnormalities
Description: Vital signs categorical summarization criteria: 1) sitting systolic blood pressure (SBP) <90 millimeters of mercury (mmHg); 2) sitting diastolic blood pressure (DBP) <50 mmHg; 3) sitting pulse rate <40 or >120 beats per minute (bpm); 4) change from baseline (increase or decrease) in sitting DBP greater than or equal to (>=) 20 mmHg; 5) change from baseline (increase or decrease) in sitting SBP >=30 mmHg.
Time Frame: From first dose of study treatment (Day 1) up to Week 16
Population: All participants who received at least 1 dose of investigational product (PF-06700841 or placebo) and had post-baseline vital signs data.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Number analyzed (Participants) | 25 | 29 | 25 | 25 | 28 | 25 | 30 | 23
Participants
  Sitting DBP <50 mm Hg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting DBP increase >=20 mm Hg | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 0
  Sitting DBP decrease >=20 mm Hg | 3 | 0 | 2 | 2 | 1 | 2 | 2 | 1
  Sitting SBP <90 mm Hg | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting SBP increase >=30 mm Hg | 1 | 3 | 2 | 1 | 0 | 1 | 0 | 0
  Sitting SBP decrease >=30 mm Hg | 2 | 2 | 1 | 2 | 1 | 3 | 2 | 1
  Sitting pulse rate <40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting pulse rate >120 bpm | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

14. Secondary Outcome: Number of Participants With Post-Baseline Electrocardiogram (ECG) Abnormalities
Description: ECG categorical summarization criteria: 1) QRS duration (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization): >=140 milliseconds (msec), >=50% change from baseline; 2) PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization): >=300 msec, >=25% change when baseline is > 200 msec or >=50% change when baseline is less than or equal to (<=) 200 msec; 3) QT interval (time from ECG Q wave to the end of the T wave corresponding to electrical systole): absolute value of >=500 msec; 4) QTc interval (QT corrected for heart rate): absolute value of 450 to <480 msec, 480 to <500 msec, >=500 msec; a change from baseline of 30 to <60 msec or >=60 msec.
Time Frame: From first dose of study treatment (Day 1) up to Week 16
Population: All participants who received at least 1 dose of investigational product (PF-06700841 or placebo) and had post-baseline ECG data.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
Number analyzed (Participants) | 24 | 29 | 25 | 25 | 28 | 25 | 28 | 22
Participants
  PR interval >=300 msec | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  %Change in PR interval >=25/50% | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  QRS duration >=140 msec | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  %Change in QRS duration >=50% | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  QT interval >=500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTc >=450 to <480 msec | 6 | 1 | 2 | 0 | 1 | 1 | 0 | 1
  QTc >=480 to <500 msec | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  QTc >=500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTc change >=30 to <60 msec | 2 | 0 | 2 | 1 | 3 | 3 | 0 | 1
  QTc change >=60 msec | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 20 weeks
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD | PF-06700841 60 mg QD Followed by 10 mg QD | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) | PF-06700841 60 mg QD Followed by Placebo | PF-06700841 30 mg QD | PF-06700841 30 mg QD Followed by 10 mg QD | PF-06700841 30 mg QD Followed by 100 mg QW | Placebo
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/29 | 0/26 | 0/25 | 0/29 | 0/25 | 0/30 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/25 | 1/29 | 1/26 | 1/25 | 0/29 | 0/25 | 0/30 | 0/23
Other Adverse Events (participants affected / at risk) | 11/25 | 14/29 | 13/26 | 13/25 | 13/29 | 12/25 | 16/30 | 9/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD (N=25) | PF-06700841 60 mg QD Followed by 10 mg QD (N=29) | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) (N=26) | PF-06700841 60 mg QD Followed by Placebo (N=25) | PF-06700841 30 mg QD (N=29) | PF-06700841 30 mg QD Followed by 10 mg QD (N=25) | PF-06700841 30 mg QD Followed by 100 mg QW (N=30) | Placebo (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-06700841 60 mg Once Daily (QD) Followed by 30 mg QD (N=25) | PF-06700841 60 mg QD Followed by 10 mg QD (N=29) | PF-06700841 60 mg QD Followed by 100 mg Once Weekly (QW) (N=26) | PF-06700841 60 mg QD Followed by Placebo (N=25) | PF-06700841 30 mg QD (N=29) | PF-06700841 30 mg QD Followed by 10 mg QD (N=25) | PF-06700841 30 mg QD Followed by 100 mg QW (N=30) | Placebo (N=23)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 4 (6) | 1 (1) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (4) | 3 (3) | 3 (3) | 5 (6) | 6 (6) | 4 (5) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT02969018/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT02969018/SAP_001.pdf